CLINICAL TRIAL: NCT04716374
Title: Clonality of Pathogenic Variants in Homologous Recombination Repair Genes in Patients With Epithelial Ovarian Cancer
Brief Title: Pathogenic Variants in Homologous Recombination Repair Genes in Patients With Epithelial Ovarian Cancer
Acronym: PaVaClO
Status: Completed | Type: Observational
Sponsor: Hellenic Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: Ovarian_ΗΕ4G/20
Record Dates: First submitted 2020-12-17; First posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2020-12

CONDITIONS: Epithelial Ovarian Cancer
Keywords: Epithelial ovarian cancer; Next Generation Sequencing (NGS); Pathogenic variants; Tumor molecular profiling; Clonality; Homologous recombination repair
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with epithelial ovarian cancer: Patients with epithelial ovarian adenocarcinoma with archival tumor tissue available for analysis were identified through the Hellenic Cooperative Oncology Group (HeCOG)'s tumor repository. Patients had received treatment at HeCOG-affiliated institutions following standard international guidelines.
  Interventions: Other: Tumor molecular profiling

INTERVENTIONS:
Other: Tumor molecular profiling — Tumor tissue processing and all NGS genotyping were performed at the Laboratory of Molecular Oncology (Hellenic Foundation for Cancer Research / AUTH). Paraffin H&E sections from the retrieved tissue blocks were centrally reviewed for tumor histology and tissue adequacy for DNA extraction and were marked for macrodissection along with tumor DNA content [(former tumor cell content (TCC%)] assessment. DNA was extracted from macrodissected tissue fragments with the QIAamp® DNA mini kit (Qiagen, Hilden, Germany), measured in a Qubit fluorometer (Thermo Fisher Scientific, Paisley, UK), and genotyped with NGS in an Ion Torrent Proton sequencer (Thermo Fisher Scientific) by using a previously published custom panel (Kotoula, Lakis et al. 2019). Following stringent variant quality filtering (Kotoula, Chatzopoulos et al. 2021), 500 tumors
  Other Names: NGS

SUMMARY:
Molecular alterations in Homologous Recombination Repair (HRR) genes have been associated with clinical benefit from chemotherapy and/or Poly (ADP-ribose) polymerase (PARP) inhibitors in patients with epithelial ovarian cancer. Therefore, the performance of tumor molecular profiling is currently recommended by international guidelines at initial diagnosis, among other reasons, for the modification of the treatment plan. The investigators' hypothesis was that tumor molecular profiling reveals additional parameters that can improve the predictive and prognostic role of the mere presence of HRR gene mutations. The study aimed to investigate the prognostic and predictive role of clonality of pathogenic variants in HRR genes and/or concurrent pathogenic variants in other clinically relevant genes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with epithelial ovarian cancer
* Received treatment at HeCOG-affiliated institutions
* Have signed informed consent
* With adequate tumor tissue for analysis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with epithelial ovarian adenocarcinoma with archival tumor tissue available for analysis were identified through the Hellenic Cooperative Oncology Group (HeCOG)'s tumor repository. Patients had received treatment at HeCOG-affiliated institutions from following standard international guidelines.
  In total, 501 patients with ovarian adenocarcinoma were included in the study (median age at ovarian cancer diagnosis was 58 years). Tumor histological types included predominantly high-grade serous, followed by endometrioid and clear cell carcinomas. All except 3 patients underwent surgery at initial diagnosis, most commonly total abdominal hysterectomy with bilateral salpingo-oophorectomy.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Actual)
Dates: Start 2004-01 (Actual); Primary Completion 2013-01 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Overall survival | Through study completion, an average of 3 years
  The time from ovarian cancer diagnosis to the date of death from any cause

SECONDARY OUTCOMES:
Progression-free survival | From date of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 96 months
  The time from initiation of first-line chemotherapy to the first documented progression, death from any cause or last contact, whichever occurred first

CONTACTS AND LOCATIONS:
Overall Officials: ELENA FOUNTZILAS, MD, Principal Investigator — HeCOG

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fountzilas E, Kotoula V, Koliou GA, Liontos M, Papadopoulou K, Giannoulatou E, Papanikolaou A, Tikas I, Chrisafi S, Mauri D, Chatzopoulos K, Fostira F, Pectasides D, Oikonomopoulos G, Aivazi D, Andrikopoulou A, Visvikis A, Aravantinos G, Zagouri F, Fountzilas G. Tumor Genotyping and Homologous Recombination Repair Gene Variants in Patients With Epithelial Ovarian Cancer: Is Pathogenic Enough? Front Oncol. 2021 Jun 1;11:683057. doi: 10.3389/fonc.2021.683057. eCollection 2021. PMID 34141624